CLINICAL TRIAL: NCT07101757
Title: Neonatal Neurodevelopmental Outcomes: Addressing Family Needs and Strengthening the Caregiver-Baby Bond
Brief Title: Neonatal Neurodevelopmental Outcomes
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Episcopal Health Foundation (Unknown)
Responsible Party: Principal Investigator, Michelle Lopez, Associate Professor of Pediatrics, Baylor College of Medicine
Other Study IDs: H-57296
Record Dates: First submitted 2025-07-18; First posted 2025-08-03 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Food Insecurity; Depression; Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive Screens: * Enrollment survey
  * Referral to behavior health clinician (BHC)
  * Referral to emergency psychiatric services
  * Referral the Houston Food Bank (HFB)
  * Follow-up surveys
- Negative Screens: -Enrollment survey

SUMMARY:
The main goal of this research is to help mothers with depression and anxiety to cope and bond with their baby.

The next goal is to provide resources to help with household needs like food, rent, or utility assistance, health insurance. Our theory is that helping with food insecurity, household needs, and emotional health will help children and families.

DETAILED DESCRIPTION:
The purpose of this study is to support families of children who are hospitalized. Participants will be asked to complete a survey regarding resources that may enhance caregiver wellbeing. These resources are intended to also support the health and developmental potential of the hospitalized child.

There is a small risk of loss of confidentiality associated with participation in the research; however, the investigators have implemented multiple safeguards to protect participant information. There is no guarantee of direct benefit from participation. If a need for resources is identified, participants may be referred to hospital-based food resources or a local food bank, which could be beneficial.

Additionally, many mothers of hospitalized children experience symptoms of depression, anxiety, and stress. A program is available within the hospital that includes access to a specialist and supportive resources for those experiencing such feelings.

The findings from this study may inform future efforts to assist caregivers more effectively. Participation in this research is voluntary, and individuals may instead request a social work consultation to determine eligibility for available resources without enrolling in the study.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of young infants (0-6 months of age) hospitalized at Texas Children's Hospital intensive care or acute care units.
* English or Spanish speaking caregiver.
* Age of caregiver ≥ 18 years old.
* Caregiver willing to complete study procedures.

Exclusion Criteria:

* Caregivers who do not have primary custody.
* Caregivers who live outside of Texas (due to lack of Houston Food Bank resources outside of Texas).
* Children in CPS custody.
* Caregiver is not the primary caregiver.
* Previous enrollment in this study.
* Neonates who are non-viable

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include adult caregivers (18 years or older) who speak English or Spanish and have infants aged 0-6 months hospitalized at Texas Children's Hospital. Caregivers must be willing to participate in study activities. Those without primary custody, living outside Texas, or previously enrolled in the study will not be eligible
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Implementation | 12 months
  Assessed by the proportion of eligible participants who enroll and complete the intervention protocol.
  Unit of Measure: Percentage of participants completing the intervention.
Acceptability of Intervention | 12 months
  Measured using the Acceptability of Intervention Measure (AIM), a validated 4-item Likert scale assessing participant perceptions of the intervention.
  Unit of Measure: Mean AIM score (range: 1-5).
Caregiver Mental Health Outcomes | 12 months
  Evaluated using the Patient Health Questionnaire-9 (PHQ-9) for depression and the Generalized Anxiety Disorder-7 (GAD-7) scale for anxiety.
  Unit of Measure: Mean scores on PHQ-9 and GAD-7.
Caregiver-Infant Bonding and Nurture | 12 months
  Assessed using the Postpartum Bonding Questionnaire (PBQ) to evaluate caregiver-infant bonding.
  Unit of Measure: Mean PBQ score.
Addressing Non-Medical Drivers of Health | 12 months
  Measured by the number of referrals made to food, housing, or mental health resources and the proportion of participants who accessed at least one referred service.
  Unit of Measure: Count of referrals and percentage of participants accessing services.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared with other researchers.